CLINICAL TRIAL: NCT04812600
Title: Microfluidic-based Tactile Sensor for Arterial Pulse Signal Measurements in Patients Going Through Cardiac Rehabilitation
Brief Title: Microfluidic-based Tactile Sensor in Cardiac Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhili hao (Other)
Collaborators: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor-Investigator, Zhili hao, Professor, Old Dominion University
Organization: Old Dominion University (Other)
Other Study IDs: 19-04-FB-0100
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases; Vascular Stiffness; Endothelial Dysfunction
Keywords: Exercise; vascular disease; cardiac rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Rehabilitation: Individuals assigned to phase II (outpatient) cardiac rehabilitation program will undergo their normal exercise routines while the investigators make the measurements pre and post exercise at 0 week, and following 1 and 4 weeks of exercise.

SUMMARY:
This study will examine the impact of cardiac rehabilitation on blood vessel health using a newly developed microfluidic-based tactile sensor to assess blood vessel health. The participants will have their blood vessel health measured using a sensor that is placed on top of the skin over the artery before and after exercise (1, 3, 5, 10, 30 and 60 mins). The investigators will study these responses at the first session of cardiac rehabilitation and following 1 and 4 weeks of cardiac rehabilitation (sessions 3 and 6). The investigators will also collect some information from the medical record regarding: age, gender, body mass index, resting cardiovascular measures (heart rate, blood pressure etc), medications, reasons which qualified the participant into cardiac rehabilitation, blood tests related to heart or cardiovascular function, metabolic panel, lipid panel, echocardiogram results, recorded electrocardiogram, known vascular diseases, presence of implantable devices, Seattle Heart Failure Model data and cardiovascular measures and exercise workloads during cardiac rehabilitation.

DETAILED DESCRIPTION:
The investigators will make the following research measurements (pre-exercise measurement and post-exercise measurement) on the first day of cardiac rehab, and following 1 and 4 weeks of cardiac rehabilitation.

Subjects will have their arterial pulse measured at the radial (wrist), carotid (neck) and temple (side of the head) arteries. The sensor will remain in place for 2-3 minutes while the recordings are made. Light pressure will be applied during this time. Blood pressure will also be obtained in the opposite arm.

The subject will then exercise on the modalities, intensity and duration designated by the staff in the Sentara Heart Hospital Cardiac Rehabilitation. It's important to note, that the normal standard of care will not change by the individual participating in this research study. The participants will follow standard physician ordered cardiac rehabilitation. The order of the modalities performed will be completed in the same order on the day of research testing in weeks 1 and 4.

After finishing the exercise, the subject will sit down for 1hr. The participant's pulse signals will be measured at 0-5min, 10min, 20 min, 30min and 1hr after exercise. Blood pressure will also be obtained from the opposite arm at the same time intervals.

The investigators will be collecting cardiac rehab data from each research day. This data will be entered into Redcap by the Sentara researchers.

The investigators will record from the most recent values/visits prior to start of cardiac rehab therapy, and this information will be entered into Redcap by the Sentara researchers.

The investigators will document at 1, 2 and 3 years from start of cardiac rehab, as to patient survival status.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-70
* Subjects who qualify for cardiac rehabilitation via doctor's orders

Exclusion Criteria:

●Physical limitations which would preclude one from performing exercise.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are undergoing Phase II (outpatient) cardiac rehabilitation at Sentara Heart Hospital (Norfolk, Va) and meet the inclusion and exclusion criteria listed will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-03-20 (Estimated); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
Micro-tactile sensor assessment of arterial stiffness change to exercise | The change of up to 1 hour post exercise relative to pre-exercise, at 0 weeks, 1 week and 4 weeks of cardiac rehabilitation
  Elasticity (unit measure: pascal) of arterial wall will be assessed.
Micro-tactile sensor assessment of arterial viscosity change to exercise | The change of up to 1 hour post exercise relative to pre-exercise, at 0 weeks, 1 week and 4 weeks of cardiac rehabilitation
  Damping (unit measure: pascal x sec) of the arterial wall will be assessed.
Micro-tactile sensor assessment of arterial radius change to exercise | The change of up to 1 hour post exercise relative to pre-exercise, at 0 weeks, 1 week and 4 weeks of cardiac rehabilitation
  Size of the artery lumen (unit measure: mm) will be assessed.
Automated blood pressure device assessment of systolic and diastolic blood pressure change to exercise | The change of up to 1 hour post exercise relative to pre-exercise, at 0 weeks, 1 week and 4 weeks of cardiac rehabilitation
  Systolic and diastolic blood pressure (unit measure: mmHg) of the artery will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Hao, Ph.D., Principal Investigator — Old Dominion University
Locations (1):
- Sentara Heart Hospital, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No